CLINICAL TRIAL: NCT03200626
Title: A Prospective, Multicenter, Observational Study to Evaluate Hematopoietic Progenitor Cell Mobilization in Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Observational Study to Evaluate Hematopoietic Progenitor Cell Mobilization in Patients With Newly Diagnosed Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Mehdi Hamadani, Associate Professor, Medical College of Wisconsin
Other Study IDs: SC15-04
Record Dates: First submitted 2017-06-12; First posted 2017-06-27 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Multiple Myeloma; Bone Marrow Transplant Complications
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cytokine alone or JIT plerixafor based mobilization
  Interventions: Procedure: Autologous hematopoietic cell transplant
- Routine plerixafor based mobilization
  Interventions: Procedure: Autologous hematopoietic cell transplant
- Chemomobilization
  Interventions: Procedure: Autologous hematopoietic cell transplant

INTERVENTIONS:
Procedure: Autologous hematopoietic cell transplant — Autologous hematopoietic cell transplant

SUMMARY:
Prospective, multicenter, observational registry of myeloma patients undergoing hematopoietic progenitor cell mobilization for upfront autologous transplantation.

DETAILED DESCRIPTION:
High dose therapy (HDT) and autologous hematopoietic cell transplantation (autoHCT) is considered standard therapy for younger, transplant eligible multiple myeloma (MM) patients. Mobilization of peripheral blood progenitor cells (PBPC) for HDT and autoHCT can be accomplished by using cytokines, most commonly granulocyte-colony stimulating factor (G-CSF), either alone or in combination with chemotherapy or plerixafor.

Limitations of cytokine-only mobilization in myeloma:

There is little consensus about the optimal method for PBPC mobilization in patients with MM, although there is a growing recognition of suboptimal mobilization outcomes of certain subgroups of myeloma patients mobilized with G-CSF alone. Within this context, the adverse impact of prior lenalidomide therapy on PBPC mobilization is well documented; with up to 40% of MM patients treated with lenalidomide-based induction chemotherapies not collecting ≥2 x 106 CD34+ cells/kg when mobilized with G-CSF alone.

Chemomobilization in myeloma:

In contrast, mobilization with chemotherapy (mostly cyclophosphamide) in addition to G-CSF has been shown to improve PBPC collection yield and reduce mobilization failure rates in comparison to G-CSF alone. Limited retrospective data suggest that cyclophosphamide may overcome the effects of prior lenalidomide exposure on PBPC mobilization in MM patients. Cyclophosphamide doses employed for mobilization of PBPC in MM patients in most reports have ranged from 1 gm/m2 up to 7 gm/m2. Several studies have assessed the relative impact of cyclophosphamide dose-intensity on PBPC mobilization in myeloma patients treated with conventional chemotherapy regimens. In general PBPC mobilization with high-dose cyclophosphamide (HD-CY) (7 gm/m2) plus G-CSF was found to be significantly more toxic, when compared to intermediate-dose cyclophosphamide (ID-CY) (3-4 gm/m2) and G-CSF, without any convincing evidence of superior efficacy. Studies comparing mobilization with ID-CY plus G-CSF with low-dose cyclophosphamide (LD-CY) (1-2 gm/m2) plus G-CSF, reported higher total CD34+ cell yield with ID-CY, but at the cost of higher toxicity. However, no significant difference in mobilization failure rates between the ID- and LD-CY mobilization has been reported. But these data might not be applicable to MM treated in the era of novel agents. Hamadani et al. compared the efficacy and toxicity of PBPC mobilization with G-CSF and either ID-CY or LD-CY, in MM patients receiving only novel induction regimens, and reported a more robust PBPC mobilization and significantly reduced the rates of mobilization failure with ID-CY in MM patients receiving modern inductions. Within the context of stem cell mobilization in MM patients treated with novel inductions, it appears that ID-CY and G-CSF may have a favorable risk/benefit ratio and can be considered a regimen with an optimal dose-intensity in order to assess the efficacy of novel mobilization regimens against cyclophosphamide-based mobilizing strategies. But these single center observations merit confirmation in large, multicenter datasets.

Plerixafor-based mobilization in myeloma:

Plerixafor is a small molecule that inhibits chemokine stromal cell derived factor 1-alpha from binding to CXC chemokine receptor 4, resulting in increased hematopoietic stem and progenitor cell migration into peripheral blood circulation. Plerixafor use in combination with G-CSF has resulted in significant improvements in the mobilization outcomes of MM patients. Despite the promising results of plerixafor and G-CSF for PBPC mobilization, the use of chemotherapy-based mobilization regimens remain standard practice in many transplant centers, driven in part due the costs associated with plerixafor based strategies.

Chemomobilization vs. Plerixafor-based mobilization in myeloma:

No randomized trials comparing chemomobilization vs. plerixafor plus G-CSF in patients with myeloma have been published. While a few retrospective studies have reported on the relative efficacy of cyclophosphamide-based mobilization against plerixafor and G-CSF, they included patients receiving either LD-CY or doses above 4mg/m2, contained patients with non-Hodgkin lymphoma (NHL), and likely included MM patients receiving conventional induction regimens. Awan et al. retrospectively compared that efficacy, toxicity and cost of PBPC mobilization with G-CSF and either ID-CY or plerixafor, in MM patients receiving only novel induction regimens. Compared to plerixafor, ID-CY use was associated with higher median peak peripheral blood CD34+ cell count (68/µL vs. 160/µL, p<0.001), and CD34+ cell yield on day 1 of collection (6.9 x 106/kg vs. 11.7 x 106/kg, p=<0.001). No patients in either group had mobilization failure. The total CD34+ cell yield was significantly higher in the ID-CY patients (median collection 16.6 x 106 cells/kg vs. 11.6 x 106 cells/kg; p-value <0.001). Mobilization with ID-CY was associated with significantly more frequent episodes of febrile neutropenia (16.3% vs. 0%; p=0.02), higher use of intravenous antibiotics (16.3% vs. 3%; p=0.03), transfusion support and need for hospitalizations (p=0.02). The average total cost of mobilization in the plerixafor group was significantly higher compared to the ID-CY group ($28,980 vs. $22,504.8; p-value=0.001). This study showed lower mobilization costs but greater toxicity with chemotherapy based mobilization in MM. The limitations of the analysis include small sample size and retrospective nature. Of note LD-CY in a different study was shown to be inferior to plerixafor in terms of PBPC mobilization efficacy and collection failure rates.

As needed or Just-in-time Plerixafor:

As noted previously, plerixafor combined with G-CSF provides superior mobilization outcomes in MM and NHL compared to G-CSF alone. It has also been shown to be an effective salvage option for patients failing to collect adequate CD34+ cells with G-CSF alone or chemomobilization [24-26]. However, the high cost of plerixafor has limited its routine use in HPC mobilization. Risk-adapted algorithms have been developed in several institutions to rescue patients at high-risk for mobilization failure and restrict plerixafor use to curtail mobilization costs. Veltri et al. recently reported a single institution comparative analysis of patients with MM and lymphoma who underwent G-CSF mobilization, with plerixafor used either routinely or as needed in patients at risk for mobilization failure. This analysis showed no mobilization failure events with either administering plerixafor routinely to all patients vs. by using a JIT approach, but showed that JIT method was associated with significantly lower collection costs.

While it is clear that PBPC mobilization has been a subject of several reports, including a recent registry analysis, these reports are limited by their retrospective nature, small sample size, heterogeneity of patient population and often missing information on healthcare resource utilization. In the current large, multicenter, observational study the investigators intend to collect detailed information regarding patient, disease, mobilization and healthcare utilization characteristic in a prospective fashion. This prospective, mobilization, registry dataset would then be used to evaluate efficacy of various mobilization regimens, their cost, associated healthcare resource utilization and impact on post transplantation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Myeloma patients ages 18-70 years.
* Undergoing upfront autoHCT (≤12 months from start of initial therapy for myeloma).

Exclusion Criteria:

* Patients with light chain (AL) amyloidosis or myeloma with associated AL amyloidosis.
* POEMS syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be reported consecutively from CIBMTR centers with comprehensive report form (CRF) level reporting. The centers will be chosen based on MM autoHCT volume, center practices for mobilization in order to ensure a fair distribution of various mobilization strategies. A total of 750 patients will be enrolled prospectively from approximately 20 selected centers.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Total CD34+ cell yield on the first apheresis | 6/1/17-1/1/19
  Evaluate efficacy of PBPC mobilization and collection in myeloma patients undergoing cytokine-only vs. chemomobilization vs. plerixafor-based mobilization efficacy parameters including total CD34+ cell yield on the first apheresis (per kg patient weight)
CD34+ cell yield | 6/1/17-1/1/19
  Evaluate efficacy parameters including total CD34+ cell yield
Number of apheresis sessions | 6/1/17-1/1/19
  Evaluate efficacy parameters including total number of apheresis sessions (comparison of means across groups)
Mobilization failure rates | 6/1/17-1/1/19
  Evaluate efficacy parameters including mobilization failure rates (defined as failure to collect ≥2 million CD34+ cells per kg patient weight)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for International Blood and Marrow Transplant Research, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
No IPD to be shared